CLINICAL TRIAL: NCT03841799
Title: COLON-IM : Prospective Cohort Study About Colorectal Environment : Microbiota and Immune Infiltrate in Normal, Dysplastic and Neoplastic Colorectal Tissue
Brief Title: COLON-IM : Microbiota and Immune Infiltrate in Normal, Dysplastic and Neoplastic Colorectal Tissue
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET18-276 (COLON-IM)
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
Keywords: Microbiota; Microenvironment colorectal tissue; Immune infiltrate
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample at surgery (no additional needle-sticks). Stool samples at surgery, at Month 3 post surgery and at Month 6 post surgery. Colorectal tissue sample from surgical specimen (healthy tissue, polyp(s), colorectal tumor).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of COLON-IM is to describe colorectal tissue microenvironment (neutrophils infiltrate) of patients with benign or malignant colorectal lesion (from stage I to III according to Tumor Node Metastasis (TNM)/ Union for International Cancer Control (UICC) classification).

DETAILED DESCRIPTION:
Colorectal cancers (CRC) are the most common gastrointestinal cancers in Western countries (both Europe and the US) ; they are both associated with significant morbidity and mortality. The 5-year survival is around 63.5% (including all stages). Sporadic colon cancers make up 85% of all colorectal adenocarcinoma. Preneoplastic lesions accumulate alterations in genes that regulate cell growth.

Patients suffering from CRC have a modified intestinal flora compared to healthy people. A specified microbiota profiled combined to genetic and immunological characteristics should be involved in colorectal carcinogenesis. Recent data have showed that responses to immunotherapies are associated with presence of certain bacteria in intestinal flora which potentially boost immune antitumor response.

Immunotherapy is highly efficient in tumors with high mutation load and Microsatellite Instability-High (MSI-H). MSI-H tumors represent 15% of local colorectal tumors. Today, it is important to understand all immune agents roles in colorectal carcinogenesis in order to describe new interesting immune checkpoints to target.

Tumor cells and tissues can escape immune surveillance and immune defense by several mechanisms. All immune cells subtypes present in the tumor, at the invasive tumor front and/or in tertiary lymphoid structures constitute the "immune context". The immune microenvironment has been shown to play a crucial role in disease progression, maintenance and resistance to therapy. All immune cells could play a pro-tumor or an anti-tumor role. For example, lymphocyte infiltrate is described as a prognostic factor in colorectal cancer : a tool (Immunoscore) has been validated as prognostic tool and it provides independent and superior prognostic value to TNM classification. This immune classification measures the host immune response at the tumor site and helps to guide treatment strategies.

Adaptative immunity is well known ; however, innate immunity should also play an early role during carcinogenesis. Role of neutrophils in the tumor microenvironment remains controversial, with evidence for both pro- and anti-tumor roles.Tumour-associated neutrophils (TANS) have an antitumorigenic in early stage of carcinogenesis or a protumorigenic functions in metastatic stage. Evidences indicate that neutrophils manifest functional plasticity during oncogenic process. Neutrophil-to-lymphocyte ratio is associated with patient prognosis ; a high ratio seems to be associated with poor prognostic.

Intestinal microbiota and immune infiltrate play key roles in colorectal microenvironment. Their interdependent interaction and their impacts on colorectal neoplasia and treatments are not well known. The primary objective of COLON-IM is to describe colorectal tissue microenvironment of patients with benign or malignant colorectal lesion (from stage I to III according to TNM/UICC classification).

ELIGIBILITY:
Inclusion Criteria:

* I1. Male or female patient 18 age or older at time of inform consent signature.
* I2. Patient Cohort A : with benign or malignant colorectal lesion (from stage I to III according to TNM/UICC classification) eligible to surgery, not previously be treated with an anticancer systemic agent (any type) and not be previously exposed to radiotherapy.

Cohort B : with localised colon/rectume adenocarcinoma, eligible to surgery, and treated by radiotherapy and/or pre-operative chemotherapy

* I3. Patient should be able and willing to comply with procedures as per protocol.
* I4. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed.
* I5. Patient must be covered by a medical insurance.

Exclusion Criteria:

* E1. Pregnant or breast-feeding female patient.
* E2. Prior treatment with : Any immunomodulatory treatment (streroids, immunosuppressive therapies) within 4 weeks prior inclusion, Any antibiotics within 8 weeks prior inclusion.
* E3. Patients with secondary malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints and is approved by the sponsor. Examples of the latter include: in-situ carcinoma of the cervix treated adequately, basal or squamous cell carcinoma of the skin. Patients previously treated for another cancer type and without evidence of relapse for at least 1 year are eligible.
* E4. Patient with inflammatory disease or autoimmune disease.
* E5. Patient under curatorship, guardianship or judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A : with benign or malignant colorectal lesion (from stage I to III according toTNM/UICC classification) eligible to surgery, not previously be treated with an anticancer systemic agent (any type) and not be previously exposed to radiotherapy.
  Cohort B : with localised colon/rectume adenocarcinoma, eligible to surgery, and treated by radiotherapy and/or pre-operative chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of colorectal tissue microenvironment of patients with locally colorectal neoplasia. | At surgery
  Rate of immune infiltrate in colorectal tissue

SECONDARY OUTCOMES:
Transcriptome profiling by RNAseq of neutrophils associated with neoplastic and preneoplastic lesions. | At surgery
  mRNA level by RNAseq from neutrophils at different preneoplastic and neoplastic stages.
Characterization of lymphocyte cells infiltrate in colorectal tissue (normal, neoplastic and preneoplastic). | At surgery
  Rate of lymphocyte cells in colorectal tissue (normal, neoplastic and preneoplastic).
Evaluation of the correlation between immune infiltrate and clinical data, microsatellite status and clinical evolution. | At surgery and through study completion, at least 42 months
  Correlation between immune infiltrate (including neutrophils infiltrate) and clinical data (neoplastic lesion stage according to TNM/UICC classification and preneoplastic lesion (low or high dysplasia), microsatellite status, clinical outcome (survival without relapse and overall survival).
Evaluation of cytokinic environment associated to neoplastic and preneoplastic lesions and evaluation of the correlation between cytokinic environment and clinical data, microsatellite status and clinical evolution. | At surgery and through study completion, at least 42 months
  Correlation between cytokinic environment and clinical data (neoplastic lesion stage according to TNM/UICC classification and preneoplastic lesion (low or high dysplasia), microsatellite status, clinical outcome (survival without relapse and overall survival)
Identification of microbiota modifications in stools and mucosa during colic carcinogenesis | At surgery, at Month 6 post-surgery, at Month 9 post-surgery
  Sequences of the variable portions of the 16s ribosomal RNA gene
Identification of potential molecular abnormalities in cancer cells from colorectal tissue and from blood samples. | At surgery
  Circulating tumor DNA and tumor DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu SARABI, Dr, Principal Investigator — Centre Leon Berard
Locations (3):
- France (3):
  - Hopital Saint Joseph Saint Luc, Lyon, Lyon
  - Clinique de L'Infirmerie Protestante, Lyon
  - Centre Leon Berard, Lyon